CLINICAL TRIAL: NCT04108260
Title: The Effectiveness of Recombinant Fusion Protein Linking Coagulation Factor IX With Recombinant Albumin (rIX-FP) in Severe Hemophilia B Patients Switching From Previous Factor IX Treatment
Brief Title: The Effectiveness of Recombinant Coagulation Factor IX With Recombinant Albumin (rIX-FP) in Severe Hemophilia B Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201907004MIPB
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Hemophilia
MeSH Terms: conditions — Hemophilia A | interventions — albutrepenonacog alfa

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm_Idelvion treated (Experimental)
  Interventions: Drug: Albutrepenonacog Alfa 1 UNT [IDELVION]

INTERVENTIONS:
Drug: Albutrepenonacog Alfa 1 UNT [IDELVION] — Clinical data will be collected from patients who suffered from hemophilia B, and switch from other FIX products to Idelvion as prophylaxis, prevention of bleeding (e.g. surgery) or treatment of bleeding.

SUMMARY:
The pivotal clinical data support prolonged dosing intervals of up to 14 days for routine prophylaxis in hemophilia B patients. The majority of adult and pediatric patients using Idelvion for routine prophylaxis had a median annualized spontaneous bleeding rate (AsBR) of 0.00. The majority (99%) of bleeding episodes were managed successfully with one or two infusions, and 94% of bleeds were controlled with only one infusion regardless of the cause or location.

The rationale for this study is to collect the effectiveness and safety data of severe hemophilia B patients treated with Idelvion following institutional standard of care. It is the aim of this study to extend the results of the clinical trial program to a broader hemophilia B population, and to compare with current alternative factor IX treatments in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with age ≥ 20 years old
* Endogenous FIX activity ≤1 IU/dL,
* At least 50 exposure days (EDs) with FIX products,
* No detectable inhibitor to FIX or inhibitor history,
* Had a minimum of 2 nontrauma-induced bleeding episodes (any type or location) treated in the 6 months preceding study entry,
* The patient or patient's parents or legal authorized representative, as applicable, are capable to understand the study objectives and procedure, and sign the written consent,
* Accept that the supply of Idelvion might be stopped once the study is completed,
* Able to complete a diary during 12 months or 50 EDs, whichever comes first.

Exclusion Criteria:

* Currently participating in an interventional clinical trial,
* Known hypersensitivity to any FIX product or hamster protein,
* Known inhibitor to FIX or inhibitor history,
* With other comorbidities which are not suitable for this study, at investigator's discretion,
* Not able to compliant with the prophylactic treatment,
* Lacking previous treatment and bleeding records.

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2020-04-21 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
AsBR | 12 months
  To evaluate AsBR of Idelvion in routine patient care

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No